CLINICAL TRIAL: NCT02285088
Title: A Phase I Randomised, Placebo-controlled, Double-blind, Single and Multiple Ascending Dose Study of the Tolerability and Pharmacokinetics of GBT440 in Healthy Subjects and Patients With Sickle Cell Disease
Brief Title: A Study of the Safety, Blood Levels and Biological Effects of GBT440 in Healthy Subjects and Subjects With Sickle Cell Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Blood Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GBT440-001; 2014-003555-62 (EudraCT Number)
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Healthy Subjects; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — voxelotor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- GBT440 (Experimental): Subjects randomized 6:2 to receive daily oral dosing of GBT440 or placebo for 1 day (single dose) and up to 118 days (multiple dose)
  Interventions: Drug: GBT440
- Placebo (Placebo Comparator): Subjects randomized 6:2 to receive daily oral dosing of GBT440 or placebo for 1 day (single dose) and up to 118 days (multiple dose)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GBT440 — GBT440 will be administered as oral capsules
  Arms: GBT440
Drug: Placebo — Matching placebo will be administered as oral capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetic, and pharmacodynamic effects of GBT440 compared with placebo in healthy subjects and subjects with sickle cell disease (SCD).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female of non-child bearing potential; 18 to 55 years old; are non-smokers and have not used nicotine products within 3 months prior to screening.
* Male or female, 18 to 60 years old, with sickle cell disease (hemoglobin SS, HbS/β0thalassemia, HbS/β+thalassemia, or HbSC) not requiring chronic blood transfusion therapy; without hospitalization in 30 days before screening or receiving blood transfusion within 30 days before screening; subjects are allowed concomitant use of hydroxyurea if the dose has been stable for the 3 months prior to screening.

Exclusion Criteria:

* Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Subjects who consume more than 14 (female subjects) or 21 (male subjects) units of alcohol a week.
* Subjects who have used any investigational product in any clinical trial within 30 days of screening
* Subjects with sickle cell disease who smoke >10 cigarettes per day; have hemoglobin level <6 g/dL or >10.4 g/dL (> ULN (appropriately corrected for gender) for Cohort 15) at screening; have aspartate aminotransferase (AST) >4x upper limit of normal or alanine aminotransferase (ALT), or alkaline phosphatase (ALK) >3x upper limit of normal reference range (ULN) at screening; have moderate or severe renal dysfunction

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Safety, as assessed by frequency and severity of adverse events (AEs), and changes in vital signs, 12-lead electrocardiograms (ECGs), and laboratory assessments as compared to baseline | 30 - 118 days

SECONDARY OUTCOMES:
Blood and plasma area under the concentration time curve (AUC) of GBT440 | 30 - 118 days
Blood and plasma maximum concentration (Cmax) of GBT440 | 30 - 118 days
Blood and plasma time to maximum concentration (Tmax) of GBT440 | 30 - 118 days
Percentage of hemoglobin occupied or modified by GBT440 | 30 days
Change from baseline in heart rate and pulse oximetry following exercise testing in healthy volunteers | 30 days

OTHER OUTCOMES:
Percentage of sickled cells under ex vivo conditions | 30 - 90 days
Effect of GBT440 on hemolysis as measured by LDH, direct bilirubin, hemoglobin, and reticulocyte count | 30 - 118 days
Change from baseline in pain as measured by visual analog scale | 30 days
Change from baseline in fatigue as measured by questionnaire | 30 - 118 days
Exercise capacity as measured by 6-minute walk test | 30 - 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Josh Lehrer-Graiwer, MD, Study Director — Global Blood Therapeutics; Timothy Mant, FRCP FFPM, Principal Investigator — Guy's Hospital
Locations (1):
- Guy's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Howard J, Hemmaway CJ, Telfer P, Layton DM, Porter J, Awogbade M, Mant T, Gretler DD, Dufu K, Hutchaleelaha A, Patel M, Siu V, Dixon S, Landsman N, Tonda M, Lehrer-Graiwer J. A phase 1/2 ascending dose study and open-label extension study of voxelotor in patients with sickle cell disease. Blood. 2019 Apr 25;133(17):1865-1875. doi: 10.1182/blood-2018-08-868893. Epub 2019 Jan 17. PMID 30655275